CLINICAL TRIAL: NCT04867070
Title: Pain Management in Laparoscopic Living-donor Nephrectomy: The Impact of Erector Spinae Plane Block (ESPB) on Perioperative Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Bora Dinc, Assistant Professor, MD, Akdeniz University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pain management in LLDN
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Pain, Postoperative; Donor Site Complication
Keywords: pain management; laparoscopic living-donor nephrectomy; erector spinae plane block
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Intervention Model Description: After the application of the ESPB was explained to the volunteers, a block was applied if the patients provided their consent. The donors were randomly assigned to Group B (ESPB group) or Group C (control group) using computer-generated random numbers placed in separate closed envelopes that the study investigator opened before performing the block in the operation room.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LLDN with ESPB (Active Comparator): The patient will be interviewed for participation in the study, and the pain scores of the patients who will participate in the study will be recorded according to the NAS and W-BAS scores at the first, 2nd, 12th, and 24th hours. At the end of the 24th hour, analgesic consumption will be recorded.
  Interventions: Diagnostic Test: NAS score
- LLDN without ESPB (No Intervention): The patient will be interviewed for participation in the study, and the pain scores of the patients who will participate in the study will be recorded according to the NAS and W-BAS scores at the first, 2nd, 12th, and 24th hours. At the end of the 24th hour, analgesic consumption will be recorded.

INTERVENTIONS:
Diagnostic Test: NAS score — Participants will be recorded according to the NAS and W-BAS pain scores
  Other Names: W-BAS score
  Arms: LLDN with ESPB

SUMMARY:
Laparoscopic living donor nephrectomy (LLDN) is a safe procedure and rapid wound healing, affecting the quality of life. The physiology of postoperative pain after LLDN has been attributed to reasons such as tissue damage, residual pneumoperitoneum, and diaphragm irritation. In terms of patient comfort after LLDN, pain control is provided by IV analgesics, local anesthetic injection instead of incision, and regional techniques. Regional anesthesia techniques for postoperative pain control have become popular in recent years. Today, many blocks are performed with ultrasonography (USG) to reduce the severity of pain after laparoscopic and open surgeries. In 2016, Forero et al. erector spinae plane block (ESPB) had been defined and used successfully in thoracic and abdominal surgeries. In our clinic, peripheral nerve blocks such as intravenous patient-controlled analgesia (PCA) and ESPB are applied for postoperative analgesia. The method of analgesia is suitable for the surgery and explained to the patients. This study; In LLDN operations, it was aimed to compare the bilateral ESP block performed with USG in terms of postoperative pain scores and opioid analgesic consumption compared to patients without any block. Before the operation, the anesthesiologist in charge of the anesthesia outpatient clinic provides information about both anesthesia and postoperative pain management methods suitable for surgery. This is the standard practice in our clinic. Before anesthesia, anesthesia and analgesia methods will be briefly reminded to the patient who has come for the operation. He/she will be asked if he/she wants to apply postoperative analgesia. Block procedure will be applied to patients who want ESP block. Standard analgesia will be applied to all patients. Regardless of the study, patients who underwent LLDN operation will be interviewed in the postoperative period with or without an ESP block for postoperative analgesia. The data and postoperative evaluations of the patients who agreed to participate in the study will be recorded for study purposes. The patient data will be taken from the hospital registration system.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18-75 who were operated on under general anesthesia for LLDN surgery and agreed to participate in the study will be included.

Exclusion Criteria:

* Participants who did not accept the study, had intraoperative complications, and whose laparoscopic operation was canceled will not be included in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Pain score | in 24 hours
  Pain scores between the two groups will be compared

SECONDARY OUTCOMES:
The total consumption of analgesic drugs | in 24 hours
  The total consumption of analgesic drugs between the two groups will be compared

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hosgood SA, Thiyagarajan UM, Nicholson HF, Jeyapalan I, Nicholson ML. Randomized clinical trial of transversus abdominis plane block versus placebo control in live-donor nephrectomy. Transplantation. 2012 Sep 15;94(5):520-5. doi: 10.1097/TP.0b013e31825c1697. PMID 22902793
- [Background] Hacibeyoglu G, Topal A, Arican S, Kilicaslan A, Tekin A, Uzun ST. USG guided bilateral erector spinae plane block is an effective and safe postoperative analgesia method for living donor liver transplantation. J Clin Anesth. 2018 Sep;49:36-37. doi: 10.1016/j.jclinane.2018.06.003. Epub 2018 Jun 5. No abstract available. PMID 29883965
- [Background] Daghmouri MA, Akremi S, Chaouch MA, Mesbahi M, Amouri N, Jaoua H, Ben Fadhel K. Bilateral Erector Spinae Plane Block for Postoperative Analgesia in Laparoscopic Cholecystectomy: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Pain Pract. 2021 Mar;21(3):357-365. doi: 10.1111/papr.12953. Epub 2020 Oct 25. PMID 32979028